CLINICAL TRIAL: NCT01278979
Title: Diagnosing Perineal Tears. Consistency in Midwifes Clinical Judgement When Assessing Perineal Tears Using Two Different Assessment Methods.
Brief Title: Diagnosing Perineal Tears, Does Different Assessment Methods Affect the Midwife's Clinical Judgement of Perineal Tears?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Ann Morris, authorized midwife and master student, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ann2010
Record Dates: First submitted 2011-01-11; First posted 2011-01-19 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Obstetric Perineal Rupture
Keywords: obstetric; perineal tear; perineal injury; diagnosis
MeSH Terms: conditions — Disease | interventions — Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assessment of perineal tears (Active Comparator): Consenting women sustaining perineal tear after child birth
  Interventions: Device: Objective measurements of perineal tears with "Peri-Rule"
- Visual and digital assessment (Other): Consenting women that sustained perineal tear after child birth.
  Interventions: Other: Visual and digital assessment

INTERVENTIONS:
Device: Objective measurements of perineal tears with "Peri-Rule" — Four measurements will be used in this study.
  1. Depth of tear, from the fourchette into the greatest depth of the perineal body.
  2. Length of tear, from the fourchette to the apex of the vaginal tear.
  3. Length of tear, from the fourchette along perineal skin towards the anus.
  4. Length of the perineal body, from the fourchette to outer margin of anus.
  Other Names: Peri-Rule
  Arms: Assessment of perineal tears
Other: Visual and digital assessment — Midwifes assessing perineal tears as standard procedure with visual and digital examination of the perineal tear.
  Other Names: Visual assessment; Digital assessment
  Arms: Visual and digital assessment

SUMMARY:
This study aims to compare different midwife practitioners assessments of perineal tears.

DETAILED DESCRIPTION:
Perineal injuries are one of the traumas most frequently suffered by women during delivery.Countries report wide variations in trauma rates, and within countries further variations exists among institutions and also among professional groups of caregivers.Visual and digital examination of the wound has been and is the most common way to assess and classify a perineal tear. However resent studies indicate that many tears diagnosed with this method are misclassified.The suggested reasons for this, apart from the fact that bleeding and tissue oedema make the diagnose difficult, is that many healthcare providers have too little training in perineal assessment and basic anatomy.

In this prospective randomised trial consenting women will be randomised in to the common visual and digital assessment of the perineal tear by to different midwives, blinded to each others assessment or visual and digital assessment and measuring of the tear with a small soft ruler, Peri-Rule also by two different midwives.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous vaginal birth
* Women over 18 years of age
* Healthy Child
* Written consent signed by participant
* Spontaneous tear in perineum that involves the perineal skin

Exclusion Criteria:

* Bleeding from tears that demand suturing immediately.
* Bleeding that affected the general condition negatively
* Complex tears that branched out in two or more different directions
* Women delivered instrumentally forceps or ventouse
* Women delivered with Cesarian section
* Women who sustain episiotomy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To investigate how different assessment methods affected the midwives´ clinical judgement between different midwife practitioners when they classify and evaluate perineal tears. | One and a half years
  Assessment of perineal tears using different two different assessment methods

SECONDARY OUTCOMES:
Consistency between different midwife practitioners when the classify and evaluate perineal tears. | One and a half years
  Two different midwife practitioners' assess the same perineal tear and fill out an assessment protocol independently.

CONTACTS AND LOCATIONS:
Overall Officials: Ann IC Morris, Reg. Midwife, Principal Investigator — Ostfold HT
Locations (1):
- Ostfold Hospital Trust, Fredrikstad, Østfold fylke, Norway